CLINICAL TRIAL: NCT04040140
Title: Integrating Auricular Point Acupressure Into Real-world Nursing Practice to Manage Cancer-related Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to Covid 19.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00183805
Record Dates: First submitted 2019-07-30; First posted 2019-07-31 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Cancer-related Pain; Acupressure
Keywords: Auricular Point Acupressure; Cancer-related Pain; Acupressure; Nursing education
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- APA Treatment (Experimental): Oncology patients with a pain rating of four or greater will receive APA treatment for patients' cancer-related pain. The ear points will be determined by the corresponding body points related to the patient's specific pain. Pain data will be tracked by electronic surveys and Electronic Health Records.
  Interventions: Other: APA Treatment

INTERVENTIONS:
Other: APA Treatment — Light touch using vaccaria seeds on corresponding ear points related to patient's pain.

SUMMARY:
The aims of this proposal are to (1) examine the feasibility of providing a training course of Auricular Point Acupressure (APA) for clinical oncology nurses who can integrate APA into real-world nursing care settings and (2) examine the effectiveness of APA on cancer-related pain (CRP) under the usual conditions.

DETAILED DESCRIPTION:
Cancer-related pain (CRP) is considered one of the most challenging symptoms that cancer patients experience. Opioid use is the most common strategy to manage pain. However, pharmacological treatments are associated with a variety of adverse side effects, including drowsiness, constipation, dry mouth, and the potential for addiction. As a result, up to 52% of cancer patients do not receive adequate analgesic medication. The high prevalence of pain and ineffective CRP management highlight the limitations of current CRP strategies. An effective, nonpharmacological patient-managed strategy-that has potential to provide quick and low-cost pain relief without new side effects-is an essential next step to manage CRP.

Auricular point acupressure (APA), a non-invasive and nonpharmacological patient-managed strategy, can be an innovative solution for CRP. APA is derived from Chinese Medicine and is different from auricular acupuncture, which is an invasive (using needles) and passive treatment (administered by a licensed practitioner). APA is a non-invasive and active treatment for patients with pain and other symptoms. It involves needleless, acupuncture-like stimulation of ear points. Small seeds are taped on specific ear points for stimulation by patients. Once the seeds have been taped on the patient's ear by the skilled provider, the patient is able to co-manage patient's treatment at home. APA is popular in Taiwan, China, and Europe. Though its use is limited in the U.S., a limited number of clinical trials have supported APA. To achieve pain relief, the participant presses on the seeds to stimulate ear points three times daily, three minutes per time, for a total of nine minutes per day. APA provides pain relief within 1-2 minutes after ear stimulation and also sustains pain relief for one month after a 4-week APA intervention. The rapid pain relief makes APA an attractive strategy to manage CRP.

The investigators' team has conducted a series of APA studies among patients with (1) chronic low back pain, (2) aromatase inhibitor musculoskeletal symptoms (AIMSS), (3) persistent post-mastectomy pain, and (4) chemotherapy-induced neuropathy (CIN). All of the investigators' pilot studies demonstrated better than a clinically significant pain reduction (30% reduction) after 4 weeks of APA and sustained effects for 1-month. Significant plasma inflammatory changes (IL-1β, IL-2, IL-6, Tumor Necrosis Factor α, and IFNγ) were found after 4 weeks, indicating that APA may affect brain macrophage-cells resulting in inflammatory cytokines alterations, leading to sustained pain relief at 1-month follow-up. Based on these findings, the investigators believe APA would be particularly suitable to reduce CRP. More importantly, easy implementation of APA and its immediate and lasting pain relief can empower and motivate cancer patients to adhere to APA treatment and allows patients to engage other forms of pain intervention, such as maintaining and/or increasing physical activity as a by-product of improved analgesia.

Nurses are the patient's first line of support in managing CRP; however, nurses have limited tools available to accomplish this. The most common treatments that nurses have at nurses' disposal are the usage of analgesics or referrals to specialty consultations. Once patients are referred, the role of nurses as cohesive guides and caretakers is often lost. To address this dilemma, patients and nurses need access to a therapy that can quickly relieve the pain, which, in turn, reduces the analgesic use and encourages patients and nurses to engage in other pain interventions. Due to the non-invasive characteristic of APA, nurses can learn APA and incorporate it into nurses' practice to provide pain relief and augment the effects of other pain interventions.

The aims of this proposal are to (1) examine the feasibility of providing a training course of APA for clinical oncology nurses which can integrate APA into real-world nursing care settings and (2) examine the effectiveness of APA on CRP under the usual conditions.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients with worst pain rated as 4 or more on a 0-10 numeric rating scale in the last 24 hours, which will use the EPIC pain scale
* Able to read and write English
* Able to apply pressure to the seeds taped to the ears. Patients with any cancer type will be eligible for this study so long as the patients are experiencing cancer-related pain
* Owns a smartphone

Exclusion Criteria:

* Is delirious
* Has ear skin disease
* Non-English speaker
* Has latex allergy to the tape used for this study
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity as assessed by the Brief Pain Inventory (BPI) short form | Baseline (pre-treatment), APA Intervention (one session, 1 day), Follow-up (3 consecutive days after treatment, starting the first day treatment is given).
  Pain intensity in the last 24 hours (1) at its worst and (2) on average will both be measured on a scale of 0 (no pain) to 10 (pain as bad as you can imagine).
Change in Pain Interference as assessed by the Brief Pain Inventory (BPI) short form | Baseline (pre-treatment), APA Intervention (one session, 1 day), Follow-up (3 consecutive days after treatment, starting the first day treatment is given).
  Pain interference with general activity, mood, walking ability, normal work, relationships with other people, sleep and enjoyment of life will be measured on a scale of 0 (does not interfere) to 10 (completely interferes).
Change in Dose of Analgesic Use | Baseline (pre-treatment), APA Intervention (one session, 1 day), Follow-up (3 consecutive days after treatment, starting the first day treatment is given).
  Dose of analgesic use will be collected in electronic health record (EHR) as part of routine nursing assessments for patient care.

SECONDARY OUTCOMES:
Change in Fatigue as assessed by a 0 to 10 scale | Baseline (pre-treatment), APA Intervention (one session, 1 day), Follow-up (3 consecutive days after treatment, starting the first day treatment is given).
  Fatigue will be measured on a scale of 0 (energetic, no fatigue) to 10 (worst possible fatigue).
Change in Quality of Sleep as assessed by a 0 to 10 scale | Baseline (pre-treatment), APA Intervention (one session, 1 day), Follow-up (3 consecutive days after treatment, starting the first day treatment is given).
  Sleep quality will be measured on a scale of 0 (very poor) to 10 (very good).

CONTACTS AND LOCATIONS:
Overall Officials: Chao Hsing Yeh, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Van de Castle B, Lukkahatai N, Billing BL, Huang X, Wu H, Zhang J, Abdi S, Kameoka J, Smith TJ. Nurse-Administered Auricular Point Acupressure for Cancer-Related Pain. Integr Cancer Ther. 2023 Jan-Dec;22:15347354231198086. doi: 10.1177/15347354231198086. PMID 37706457